A clinical prospective study to validate a risk scoring model integrated preoperative immune-inflammatory indicators, tumor markers and imaging examination for the lymph node metastasis of gastric cancer before surgery (DJY004 Trail)

**Edition Number: 1.0** 

Edition Generation Date: Jul 01, 2023 Principal Investigator: Jingyu Deng

Research Institute: Cancer Hospital & Institute of Tianjin Medical University

## **Protocol:**

- Curative gastrectomy and D2 lymphadenectomy
- Postoperative pathology confirmed gastric cancer without distant metastasis or peritoneal dissemination (M0)
- Age between 18 and 70 years
- KPS score >60
- No autoimmune, inflammatory, or blood diseases, no active infection
- No seriously chronic diseases of important organs
- No other malignancies

Patients included in the study

N>100

on of preoperative clinical data of patients including:

Collection of preoperative clinical data of patients including: CT examination results (regional lymph nodes with a maximum short diameter ≥10mm considered positive), PLR, CEA, CA242, CA724 levels.

Calculation of lymph node metastasis risk of patients based on the previously constructed prediction model.

Collection of postoperative pathological data and lymph node status of patients.

To analyze the consistency between the actual results of postoperative lymph node metastasis occurrence and the predicted results by the risk scoring model to identify the clinical applicability of the model.